CLINICAL TRIAL: NCT03199677
Title: An Exploratory Single-center, Open-label , Clinical Study of Apatinib in Patients With Local Progressive/Metastatic Refractory Thyroid Cancer
Brief Title: A Clinical Study of Apatinib in Patients With Local Progressive/Metastatic Refractory Thyroid Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Shengyu Zhou, Deputy director of the physician, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AHEAD-RTC001
Record Dates: First submitted 2017-06-16; First posted 2017-06-27 (Actual); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Refractory Cancer
Keywords: apatinib,refractory thyroid cancer
MeSH Terms: conditions — Neoplasms; Thyroid Neoplasms | interventions — apatinib

STUDY DESIGN:
Intervention Model Description: single group,apatinib 500mg po qd,d1-28
Masking Description: no parallel,no control
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- apatinib with 500mg qd po (Experimental): Patients administrate apatinib with the dose of 500mg once per day,half an hour after a meal.
  Interventions: Drug: Apatinib

INTERVENTIONS:
Drug: Apatinib — Apatinib is an oral tyrosine kinase inhibitor.

SUMMARY:
This is a single-center, open-label, single arm，exploratory clinical trial evaluating the efficacy and safety of Apatinib in patients with local progressive/metastatic refractory thyroid cancer.

DETAILED DESCRIPTION:
This is a single-center, open-label, single arm，exploratory clinical trial evaluating the efficacy and safety of Apatinib in patients with local progressive/metastatic refractory thyroid cancer.

The primary endpoint is objective response rate(ORR),the secondary endpoints include progression-free-survival(PFS)；disease control rate(DCR);serum Tg、TgAb、calcitonin；safety.

If any case happens as following,including withdrawing informed consent form(ICF)、unbearable toxicity or adverse reactions、other conditions which investigators think the patients are unsuitable to go on trail,the patient will not go on trial any longer,or every subject will obtain study treatment until tumor progress with CT/MRI proof.The indicators of efficacy and safety will be always observed during the trail process.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years old，gender limitation.
2. The pathologic subtype of thyroid carcinoma, which was confirmed by histopathological histology, included iodine refractory thyroid papillary carcinoma and follicular carcinoma, medullary thyroid carcinoma and undifferentiated carcinoma.
3. Patients with at least one measurable lesion (RECIST1.1), at least one measurable lesion after the treatment (spiral CT scan length to diameter 10 mm or higher, according with the requirement of RESCIST version 1.1 standard).
4. Radioactive iodine deficiency (according with one of the following conditions):

   1. The target lesion was completely deprived of iodine in the treatment of radioactive iodine;
   2. The patients were treated with single dose of iodine (3.7 GBq) and the disease progressed in 12 months;
   3. The patients were given an iodine treatment interval of less than 12 months, and the dose was greater than that 3.7 GBq [≥100mCi], with at least one iodine treatment over 12 months of disease progression;
   4. Cumulative doses of radioactive iodine were greater than 22.2 GBq (or more than 600 mCi).
5. Patients who underwent at least one failure of standard chemotherapy can be recommended to get into the group.
6. Organs function have to be compliant with the following specifications:

   ANC≥1.5×109/L; PLT≥100×109/L; Hb≥90g/L; TBIL≤1.5×ULN; ALT &AST ≤2.5×ULN ; ALT &AST ≤5×ULN in patients with hepatic metastasis; BUN & Cr≤1×ULN, CCR≥50mL/min (Cockcroft-Gault formula); Normal coagulation function (INR<1.5 or PT<ULN+4s or APTT<1.5 ULN); Urinary protein<++ or urine protein quantitation in 24 hours ≤1.0 g.
7. Life expectancy ≥ 12 weeks.
8. Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0~2.
9. Pre-menopausal women must have a negative pregnancy test within 7 days before study entry and agree to use a medically acceptable method of contraception throughout the treatment periods and for at least six weeks after treatment discontinuation.
10. The subjects volunteered to participate in the study, sign informed consent forms, and compliance with follow-up.

Exclusion Criteria:

1. The presence of a third interstitial fluid (such as a large amount of pleural effusion and/or peritoneal fluid, pericardial fluid) that cannot be controlled by a drainage or other methods.
2. Before or at the same time with other malignant tumors, except cured skin basal cell carcinoma, cervical carcinoma in situ or other effective treatment of tumors and did not see signs of disease for five years.
3. The patients who used VEGFR-TKI drugs, such as Vandetanib， Cabozantinib， Lenvatinib，Sunitinib，Sorafenib in one month.
4. Inability to swallow, chronic diarrhea and obstruction of the intestine, various factors which affect drug use and absorption.
5. major surgical or severe trauma injuries, fractures, or ulcers before 4 weeks of enrolling , 3 weeks of radiation therapy (except for partial palliative radiation), chemotherapy, and molecular target therapy in three weeks, Treatment with nitrocarbamide or mitomycin before six weeks of enrolling.
6. uncontrolled hypertension (systolic blood pressure of 140mmHg or diastolic pressure is greater than 90mmHg, despite the best drug treatment).
7. Patients used to suffer from severe cardiovascular diseases: Ⅱ magnitude of myocardial ischemia and myocardial infarction, poor control of cardiac arrhythmias (including QTc interphase male ≥450ms, female≥470ms); According to NYHA standard, Ⅲ ~ Ⅳ cardiac insufficiency, or heart color indicate left ventricular ejection fraction (LVEF) < 50%.
8. History of significant hemoptysis within 2 months prior to enrollment or daily hemoptysis is up to 2.5ml;with the trend of haemorrhage or prior treatment with an angiogenesis therapy.
9. Significant clinical significance of bleeding symptoms or a definite bleeding tendency happened in three months prior to screening, such as gastrointestinal bleeding, bleeding ulcers, baseline period + + and above of defecate occult blood, or those with vasculitis, etc.
10. Active brain metastasis, cancer meningitis, Spinal cord oppressor activity of brain metastases of, cancer, spinal cord compression patients, CT or MRI examination revealed brain or soft meningeal disease (patients who completed treatment and get stable symptoms with brain metastases can be into the group in 21 days prior to screening, without symptoms of cerebral hemorrhage).
11. Imaging (CT or MRI) showed that tumor lesions were less than 5mm from the large blood vessels, or the central type of tumor that had penetrated the large blood vessels, or there is a clear pulmonary void or necrotic tumor.
12. Patients accept other anti-tumor therapies at the same time.
13. Treatment of thyroid cancer radiation was received 28 days prior to screening.
14. Participated in other clinical trials within 4 weeks.
15. Active or chronic hepatitis c and/or hepatitis b infection and other active infections (determined by the investigators).
16. History of immunodeficiency disease, including human immunodeficiency virus infect(HIV), or acquired immunodeficiency disease (AID) and Congenital immunodeficiency disease, or history of organs for transplantation.
17. Abdominal fistula, digestive tract perforation or intra-abdominal abscess happened within six months prior to screening.
18. Within 12 months before the first treatment occurs artery / venous thromboembolic events, such as cerebral vascular accident (including transient ischemic attack (TIA), hematencephalon, cerebral infarction), deep vein thrombosis and pulmonary embolism, etc. Received a powerful CYP3A4 inhibitor treatment in the first 7 days before the group, or received a powerful CYP3A4 inducer in the first 12 days before the study.
19. According to the investigator's judgment, there is serious illness to endanger the safety of patients, the completion of the study (e.g: severe diabetes, renal insufficiency).
20. A history of specific neurological or psychiatric disorders, including epilepsy or dementia.
21. Other cases that the investigator found ineligible.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-07-01 (Estimated); Primary Completion 2018-06-30 (Estimated); Study Completion 2018-06-30 (Estimated)

PRIMARY OUTCOMES:
objective response rate | 1 year
  ORR is defined as the percentage of subjects having achieved confirmed Complete Response+Partial Response as best overall response according to Response Evaluation Criteria Solid Tumors(RECIST 1.1).

SECONDARY OUTCOMES:
progression-free-survival(PFS) | 1 year
  From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 12 months.
disease control rate(DCR) | 1 year
  Investigators will assess treatment response according to Response Evaluation Criteria in Solid Tumors 1.1（RECIST1.1）.
serum Tg、TgAb、calcitonin | 1 year
  Evaluating the change of serum level of Tg，TgAb or calcitonin,assessed up to 12 months.
Adverse Events(AEs) | 1 year
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0.

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided